CLINICAL TRIAL: NCT04864405
Title: A Pragmatic Randomised, Multicentre Trial Evaluating the Dose Timing (Morning vs Evening) of Endocrine Therapy and Its Effects on Tolerability and Compliance (REaCT-CHRONO)
Brief Title: Evaluating the Dose Timing (Morning vs Evening) of Endocrine Therapy and Its Effects on Tolerability and Compliance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REaCT-CHRONO
Record Dates: First submitted 2021-04-09; First posted 2021-04-28 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Endocrine Therapy; Chronotherapy; Chronotherapeutics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning administration of endocrine therapy (Active Comparator): Administration of endocrine therapy defined as, within one hour of the patient wake up time
  Interventions: Other: Morning administration of endocrine therapy
- Evening administration of endocrine therapy (Active Comparator): Administration of endocrine therapy defined as, within one hour of the patient bed time
  Interventions: Other: Evening administration of endocrine therapy

INTERVENTIONS:
Other: Morning administration of endocrine therapy — Endocrine therapy administered within one hour of patient wake up time
  Arms: Morning administration of endocrine therapy
Other: Evening administration of endocrine therapy — Endocrine therapy administered within one hour of the patient bed time
  Arms: Evening administration of endocrine therapy

SUMMARY:
Endocrine therapy is an established treatment for hormone receptor-positive breast cancer, but can cause significant side effects with deterioration in quality of life. The side effects of all forms of endocrine therapy are well recognized and can lead to treatment non-persistence or non-compliance. Chronotherapy, also called chronotherapeutics, is defined as the administration of a medication in coordination with circadian rhythm in order to minimize side effects and yield a greater efficacy. The investigators propose to perform a pragmatic, multi-centre, open-label, randomized clinical trial to establish the optimal timing (morning vs. evening) of administering endocrine therapy based on side effects and benefits in early stage breast cancer patients.

DETAILED DESCRIPTION:
Endocrine therapy is an established treatment for hormone receptor-positive breast cancer, but can cause significant side effects with deterioration in quality of life. The side effects of all forms of endocrine therapy are well recognized and can lead to treatment non-persistence or non-compliance. Compliance is defined as the degree or extent of conformity to the recommended administration by the provider, whereas persistence refers to the act of continuing treatment for a certain prescribed duration. Treatment adherence is especially important in breast cancer, as early cessation or reduced compliance to hormonal therapy are associated with reduced disease-free survival and increased mortality. Chronotherapy, also called chronotherapeutics, is defined as the administration of a medication in coordination with circadian rhythm in order to minimize side effects and yield a greater efficacy. The investigators propose to perform a pragmatic, multi-centre, open-label, randomized clinical trial to establish the optimal timing (morning vs. evening) of administering endocrine therapy based on side effects and benefits in early stage breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an early stage or locally advanced hormonal receptor positive breast cancer
* Plan to receive endocrine therapy
* 18 years of age or older
* Able to provide oral consent
* Willing and able to complete questionnaires as per study protocol

Exclusion Criteria:

* Metastatic cancer
* Previous endocrine therapy for breast cancer
* Plan to receive adjuvant abemaciclib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2023-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Savard, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario

REFERENCES:
- [Background] Beltran-Bless AA, Vandermeer L, Ibrahim MFK, Hutton B, Shorr R, Savard MF, Clemons M. Does the Time of Day at Which Endocrine Therapy Is Taken Affect Breast Cancer Patient Outcomes? Curr Oncol. 2021 Jul 6;28(4):2523-2528. doi: 10.3390/curroncol28040229. PMID 34287262
- [Result] Savard MF, Ibrahim M, Saunders D, Pond GR, Ng TL, Awan AA, Sehdev S, Alqahtani N, Vandermeer L, MacDonald F, Beltran-Bless AA, Fallowfield L, Clemons M. A pragmatic, multicenter, randomized trial comparing morning versus evening dosing of adjuvant endocrine therapy (REaCT-CHRONO Study). NPJ Breast Cancer. 2025 May 29;11(1):49. doi: 10.1038/s41523-025-00762-7. PMID 40442096
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morning Administration of Endocrine Therapy | Evening Administration of Endocrine Therapy
Started | 122 | 123
Completed | 115 | 112
Not Completed | 7 | 11
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Did not want endocrine therapy | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morning Administration of Endocrine Therapy | Evening Administration of Endocrine Therapy | Total
Number analyzed (Participants) | 122 | 123 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.5) | 61.0 (11.2) | 61.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex (male/female) was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 122 | 123 | 245
Type of endocrine therapy [Count of Participants; unit: Participants] — Participants can be counted in more than one category
  Participants
    Tamoxifen | 93 | 94 | 187
    Anastrozole | 20 | 22 | 42
    Letrozole | 9 | 7 | 16
    Exemestane | 0 | 0 | 0
    LHRH | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Endocrine Toxicity and Tolerability at 12 Weeks
Description: Measured by the change in total Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) questionnaire from baseline to 12 weeks following the beginning of endocrine therapy. FACT-ES is a validated sub scale of the Functional Assessment of Chronic Illness Therapy (FACIT) measurement system. FACT-ES consists of 46 items on a 5 point Likert type scale ranging from 0 (not at all) to 4 (very much), with a total range of 0 to 184. Higher FACT-ES scores indicate better outcomes. The current outcome is a change in FACT-ES scores.
Time Frame: Baseline to 12 weeks after treatment initiation
Population: The participants who answered the FACT-ES at baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Morning Administration of Endocrine Therapy | Evening Administration of Endocrine Therapy
Number analyzed (Participants) | 103 | 102
units on a scale | -2.2 (14.1) | -5.0 (16.8)

2. Secondary Outcome: Change in Endocrine Toxicity and Tolerability
Description: Measured by the change in total score and individual Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) questionnaires from baseline to 4, 8, 12 and 52 weeks following the beginning of endocrine therapy. FACT-ES consists of 46 items on a 5 point Likert type scale ranging from 0 (not at all) to 4 (very much), with a total score range of 0 to 184. Higher scores indicate better quality of life. The current outcome is a change in FACT-ES scores over time.
Time Frame: Baseline, 4, 8, 12 and 52 weeks after treatment initiation
Population: The number analyzed differs from overall number analyzed because not all participants completed the questionnaires at all timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Morning Administration of Endocrine Therapy | Evening Administration of Endocrine Therapy
Number analyzed (Participants) | 122 | 123
units on a scale
  Baseline to 4 Weeks: number analyzed (Participants) | 106 | 108
  Baseline to 4 Weeks | -0.3 (12.6) | -0.5 (14.6)
  Baseline to 8 Weeks: number analyzed (Participants) | 105 | 104
  Baseline to 8 Weeks | -1.6 (13.7) | -2.3 (13.6)
  Baseline to 12 Weeks: number analyzed (Participants) | 103 | 102
  Baseline to 12 Weeks | -2.2 (14.1) | -5.0 (16.8)
  Baseline to 52 Weeks: number analyzed (Participants) | 102 | 101
  Baseline to 52 Weeks | -3.0 (18.7) | -4.7 (15.6)

3. Secondary Outcome: Change in Health Related Quality of Life Scores
Description: Measured by the change in the total score and individual sub scales of the validated Functional Assessment of Cancer Therapy for patients with Breast cancer (FACT-B) questionnaire from baseline to 4, 8, 12 and 52 weeks following the beginning of endocrine therapy. The FACT-B consists of 37 items on a 5 point Likert type scale ranging from 0 (not at all) to 4 (very much), with a total score range of 0 to 148. Higher FACT-B scores indicate better quality of life. The current outcome is a change in FACT-B scores over time.
Time Frame: Baseline, 4, 8, 12 and 52 weeks after treatment initiation
Population: The number analyzed differs from the overall number of participants analyzed because not all participants completed all questionnaires at all timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Morning Administration of Endocrine Therapy | Evening Administration of Endocrine Therapy
Number analyzed (Participants) | 122 | 123
units on a scale
  Baseline to 4 Weeks: number analyzed (Participants) | 106 | 108
  Baseline to 4 Weeks | 1.9 (12.0) | 1.2 (11.6)
  Baseline to 8 Weeks: number analyzed (Participants) | 105 | 104
  Baseline to 8 Weeks | 1.4 (12.3) | 0.9 (10.7)
  Baseline to 12 Weeks: number analyzed (Participants) | 103 | 102
  Baseline to 12 Weeks | 2.3 (13.6) | -0.6 (14.1)
  Baseline to 52 weeks: number analyzed (Participants) | 102 | 101
  Baseline to 52 weeks | 1.9 (18.0) | 0.8 (14.4)

4. Secondary Outcome: Number of Participants Who Were Compliant With ET
Description: Rates of non-persistence or non-compliance with initially prescribed endocrine therapy (ET)
Time Frame: 52 weeks after treatment initiation
Population: This is the modified intention-to-treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Morning Administration of Endocrine Therapy | Evening Administration of Endocrine Therapy
Number analyzed (Participants) | 111 | 110
Participants
  Still taking ET | 103 | 100
  Still taking ET at the assigned time | 105 | 105
  No interruptions of ET greater than 7 days | 103 | 95
  Still taking ET with no interruptions greater than 7 days and no change in ET type | 88 | 84

5. Secondary Outcome: Cost-effectiveness
Description: Incremental cost-effectiveness rations (cost per one quality-adjusted life year (QALY) gained).
Time Frame: 52 weeks after treatment initiation
Reporting Status: Not Posted, anticipated posting 2026-12

6. Other Pre Specified Outcome: Rates of Non-compliance to Endocrine Therapy
Description: Comparing rates of non-compliance and non-persistence to endocrine therapy with patient age, turmour stage, chemotherapy use and type of endocrine therapy. The rates of non-compliance and rates of non-persistence will be tracked throughout the duration of the study and then compared to patient age, tumour stage, chemotherapy use and the type of endocrine therapy used.
Time Frame: 52 weeks after treatment initiation
Population: This was an exploratory analysis and it was not performed.
Arm/Group | Morning Administration of Endocrine Therapy | Evening Administration of Endocrine Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Adverse events not collected. This was a pragmatic clinical trial with two standard of care arms. The protocol did not include adverse event reporting.
Arm/Group | Morning Administration of Endocrine Therapy | Evening Administration of Endocrine Therapy
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT04864405/Prot_SAP_000.pdf